CLINICAL TRIAL: NCT03792958
Title: Phase I Study of CM082 Tablets in the Treatment of Advanced Malignant Solid Tumors: Safety, Tolerance and Pharmacokinetics
Brief Title: Study of Challenge Meditech 082 (CM082) Tablets in Patients With Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AnewPharma (Industry)
Collaborators: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CM082-CA-I-105
Record Dates: First submitted 2018-12-26; First posted 2019-01-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Advanced Malignant Solid Tumors
MeSH Terms: interventions — vorolanib

STUDY DESIGN:
Intervention Model Description: The initial dose is set at 200 mg, followed by 400 mg, 600 mg and 800 mg for dose increment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM082 (Experimental): CM082 tablet
  Interventions: Drug: CM082

INTERVENTIONS:
Drug: CM082 — CM082 tablets taken orally 200、400、600 and 800 mg (QD or BID)
  Other Names: X-82

SUMMARY:
This is a Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Oral Dosing of CM082 tablets in Chinese Patients With Advanced Malignant Solid Tumors

DETAILED DESCRIPTION:
This is a single-center、open-label and non-controlled Phase 1 study which will be conducted in two parts: part A is the dose-escalation phase; part B is dose-expansion phase. The dose-escalation phase is guided by pharmacokinetics (PK) and safety, according to the standard 3+3 dose-escalation schema. CM082 tablets are taken orally with a starting dose of 200 mg and a subsequent dose of 400, 600 and 800 mg. The way of administration is as follows: QD or BID. The primary objective of this study is to determine the maximum tolerable dose (MTD)、characteristics of dose-limited toxicity (DLT) and pharmacokinetics (PK). Secondary objectives include safety、tolerability and preliminary efficacy

ELIGIBILITY:
Inclusion Criteria:

* Age:≥18 years.
* BMI generally ranges from 18-28 (BMI=Weight (Kg)/Height (m)2)
* Patients with advanced malignant solid tumors confirmed by histological or cytological examination.
* According to Recist1.1 criteria, patients have measurable or assessable tumors, and patients with advanced malignant solid tumors who have failed to respond to previous standard treatment regimens, are unable to tolerate previous treatment regimens or lack effective treatment regimens.
* Organ function level must meet the following requirements (7 days before treatment):

  * Bone marrow: absolute neutrophil count (ANC)≥1.5^109/L, platelet (PLT)≥100^109/L, hemoglobin (HB)≥9g/dL (no blood transfusion or component blood received within 14 days before detection).
  * Liver: Serum bilirubin (TBIL) ≤1.5 * upper limit of normal (ULN) , aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 * ULN (If the patient's liver metastases, AST and ALT are allowed to be ≤ 5 * ULN) ).
  * Serum creatinine≤1.5 * ULN and endogenous creatinine clearance rate≥50mL/min. According to Cockcroft-Gault formula, Please refer to attachment 7 for details.
  * International normalized ratio (INR) and activated partial thromboplastin time (APTT)≤1.5 * ULN (This provision applies only to patients who do not receive anticoagulant treatment; for patients receiving anticoagulant treatment, anticoagulants should be used within the treatment requirements).
  * Urine protein (UP)≤1+. If UP>1+, 24-hour UP should be collected for determination, and the total amount of UP should be ≤1g.
  * FT3、FT4 and thyroid-stimulating hormone (TSH) are normal or abnormal without clinical significance（Except for advanced thyroid cancer）.
* No immunodeficiency.
* The damage causes by other treatments is restored to 1 grade (CTCAE version 4.03), except for hair loss and pigmentation; If the nutritional status is stable, the long-term toxicity that cannot be recovered is allowed to exist by the investigator'judgement.
* Expected survival time≥ 3 months.
* Eastern Cooperative Group (ECOG) Performance Status score of ≤1.
* The results of serum pregnancy test for women of childbearing age should be negative within 7 days before treatment.
* Men who are fertile or women who are likely to become pregnant must use highly effective contraceptive methods (e.g., oral contraceptives, intrauterine contraceptives, sex control or barrier contraceptives combined with spermicides ) throughout the trial and continue to use contraception for 12 months after the end of treatment.
* Patients can voluntarily sign written informed consent.

Exclusion Criteria:

-Within 4 weeks before the first use of the study drug, the patient received anti- tumor drug therapy such as chemotherapy, targeted therapy, radiotherapy, biological therapy or endocrine therapy, except for the following: Nitrous urea or mitomycin C were used within 6 weeks before the first use of the study drug; Oral fluorouracil and small molecular targeted drugs were used within 2 weeks before the first use of the study drug or within 5 half-lives (whichever is the longer); Chinese medicine with anti-cancer indications was used within 1 week before the first use of the study drug.

* Surgical treatment (except biopsy) was performed within 4 weeks before the first use of study drug.
* Patients who have participated in or are participating in any other drug/therapy clinical trial (including but not limited to the anti-tumor clinical trial) within 4 weeks before treatment, counting from the time of last administration of the last clinical trial.
* Patients who received hematopoietic stimulating factors (e.g., granulocyte colony stimulating factor (G-CSF), erythropoietin, etc.) within one week before treatment.
* Pleural or ascites with clinical symptoms and requiring symptomatic treatment.
* Patients with active pulmonary disease, interstitial pneumonia or pulmonary fibrosis.
* Having any uncontrollable clinical problems or associated risk factors, including but not limited to:

  * Poorly controlled hypertension (blood pressure persistently greater than 150/90 mmHg).
  * Left ventricular ejection fraction (LVEF)≤50%.
  * The QT interval of heart rate correction (QTc) > 450 msec (males) or 460 msec (females) ( Bazett's correction (QTcB)=QT/(RR^0.5)).
  * Patients have a clinically significant history of arrhythmia or current evidence of arrhythmia, but control of atrial fibrillation for more than 30 days before administration does not affect inclusion.
  * Patients implanted with cardiac defibrillator.
  * Poorly controlled diabetes [(fasting blood glucose should not be greater than 8.9 mmol/L after drug control) refer to CTCAE version 4.03-grade 1 of hyperglycemia].
  * Heart disease (Class III/IV congestive heart failure or cardiac block defined by the New York Heart Association).
  * Decompensated cirrhosis.
  * The following conditions occur within 6 months before treatment:

    * Deep venous thrombosis or pulmonary embolism.
    * Myocardial infarction.
    * Severe or unstable arrhythmia or angina pectoris.
    * Percutaneous Coronary Intervention, Acute Coronary Syndrome, Coronary Artery Bypass Transplantation.
    * Cerebrovascular accident, transient ischemic attack or resting limping of lower limbs.
* Patients have not yet fully recovered from previous operations.
* Patients who have taken strong inhibitors and inducers of CYP3A hepatic metabolic enzymes within 2 weeks before treatment.
* Patients also take drugs that are at risk of prolonging QTc and/or Tdp.
* Patients with a history of allergy to CM082 similar drugs (e.g., sunitinib, sorafenib, pazopanib, etc.).
* Pregnant or lactating women.
* Women/men with fertility who refuse to use contraception during the trial.
* Any uncontrollable clinical problem (such as serious mental, neurological, cardiovascular, respiratory and other system diseases) or active infection that significantly affects clinical trials.
* The patient has clinical symptoms or uncontrolled central nervous system metastasis or meningeal metastasis, which is judged by the investigator to be unsuitable for admission;
* Patients with active upper gastrointestinal ulcer or other diseases known to affect drug absorption, distribution, metabolism or clearance.
* Patients with obvious abnormal gastrointestinal function such as vomiting、 diarrhea, etc..
* Positive results of HIV or Treponema pallidum antibodies (Acceptance of Treponema pallidum antibody titer test results in a Class III Grade I hospital including research centers).
* Patients with active hepatitis B or C：

  * HBsAg or HBcAb are positive, and hepatitis B virus (HBV) DNA is detected (the results are higher than the upper limit of the normal range of the research center).
  * Hepatitis C virus (HCV) antibody test results are positive, and HCV RNA is detected (the results are higher than the upper limit of the normal range of the research center).
* Patients who have progressed after using a receptor tyrosine kinase inhibitor that targets VEGFR.
* Investigators consider that it is not appropriate for subjects to participate in this study from the perspective of clinical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerable dose (MTD) or dose to absorb saturation | From the first dose to the 28th day of administration
Dose-Limiting Toxicity | From the first dose to the 28th day of administration
  Characteristics of dose-limiting toxicity (DLT), evaluation criteria: National Cancer Institute (NCI) CTC classification (version 4.03)
Pharmacokinetic parameters | From the first dose to the 28th day of administration
  Peak concentration
Pharmacokinetic parameters | From the first dose to the 28th day of administration
  Area under the time curve of blood concentration from 0 h to the last time of blood collection
Pharmacokinetic parameters | From the first dose to the 28th day of administration
  0 to Infinite Area under Blood Drug Concentration Curve
Pharmacokinetic parameters | From the first dose to the 28th day of administration
  Peak time
Pharmacokinetic parameters | From the first dose to the 28th day of administration
  Apparent terminal elimination half-life
Pharmacokinetic parameters | From the first dose to the 28th day of administration
  Terminal elimination rate constant

SECONDARY OUTCOMES:
Objective response rate | 12 months
Disease control rate | 12 months
Progression-free survival | 12 months
Overall survival | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, M.D, Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China